CLINICAL TRIAL: NCT05320003
Title: Assessment of Balance in Patients With Pes Planus Aged 50-65, Clinically and With Static Posturography
Brief Title: Assessment of Balance in Patients With Pes Planus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Shahla ALIMADATLI, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IstanbulUC-ShahlaALIMADATLI
Record Dates: First submitted 2022-03-15; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Pes Planus; Fall Risk
Keywords: Pes planus; Ink foot analysis; Pedobarography; Computed posturography
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults with pes planus (Other): Detailed clinical examination of cases with pes planus will be performed. Inky foot analysis of both feet will be performed to confirm the diagnosis of pes planus in the subjects included in the study. Staheli arch index and Chippaux-Smirak Index will be calculated for each foot based on the footprints obtained. According to the Staheli Arc Index 1 and above, according to the Chippaux-Smirak Index 0.45 and above will be considered as pes planus, static foot pressure measurement will be performed with a pedobarography device in all cases. Peak pressure, maximum force and total foot area values will be obtained. Balance assessment of the patients will be performed with a computerized static posturography device. Individuals will be graded according to the fall index results, as low, medium and high risk. It will be determined whether there is a fall risk with the Timed Up and Go Test, which is one of the clinical balance tests.
  Interventions: Diagnostic Test: Inky foot analysis; Diagnostic Test: Evaluation of plantar pressure with pedobarography; Diagnostic Test: Balance assessment with computerized posturography

INTERVENTIONS:
Diagnostic Test: Inky foot analysis — Inky foot analysis to confirm the diagnosis of pes planus
  Other Names: Fall risk assessment with static posturography
Diagnostic Test: Evaluation of plantar pressure with pedobarography — Evaluation of plantar pressure distribution by pedobarography in individuals with pes planus
Diagnostic Test: Balance assessment with computerized posturography — Evaluation of fall risk with computerized posturography

SUMMARY:
Introduction: Pes planus is a foot deformity with increased contact of the foot with the ground as a result of the decrease or disappearance of the medial longitudinal arch of the foot. The arch of the foot creates an adaptive and flexible support for the whole body, and biomechanical changes in the foot can affect the whole body posture and balance. The results of the studies evaluating balance and plantar pressure analysis in adults with pes planus seem contradictory. The aim of this study is to evaluate fall risk and plantar pressure in adults with pes planus aged 50 -65 years

DETAILED DESCRIPTION:
Materials and Methods: 34 cases with pes planus will be included in the study. Medial longitudinal arch height of all cases will be evaluated by physical examination . Affected foot, presence of "too many toes" sign will be observed. With the fingertip rise test, it will be checked whether the pes planus is flexible or rigid.

Inky foot analysis and plantar pressure analysis will be performed in cases. Chippaux-Smirak index and Staheli arch index of all cases will be evaluated for the diagnosis of pes planus.The risk of falling will be calculated by evaluation of the balance with clinically and with posturography.

Results: Statistical analyzes in the study will be made with the NCSS (Number Cruncher Statistical System) 2007 Statistical Software (Utah, USA) package program.

In addition to descriptive statistical methods (mean, standard deviation) in the evaluation of the data, the distribution of the variables will be examined with the Shapiro - Wilk normality test, one-way analysis of variance in the comparison of the normally distributed variables, Tukey multiple comparison test in the comparison of subgroups, independent t test in the comparison of the paired groups, Chi-square test will be used in comparisons of qualitative data. Results will be evaluated at the level of significance p<0.05.

Discussion: The results will be discussed according to the recent literature. In the literature, there are conflicting results about the balance and gait of adults with pes planus. In several studies in the literature, it has been found that the risk of falling is increased in elderly individuals with pes planus. The study can contribute to the literature in this perspective.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50 years and above with pes planus according to Staheli Arch Index and Chippaux- Smirak Index

Exclusion Criteria:

* Congenital anomalies of the foot
* Prior lower extremity surgery Inflammatory arthritis
* Neuromuscular diseases
* Diseases that interfere with lower extremity circulation
* Presence of orthostatic hypotension
* Untreated visual impairment
* Neurological and vestibular diseases
* Use of drugs that can cause balance disorders (Antipsychotics, Pregabalin, etc.)

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-06 (Estimated); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-05-15 (Estimated)

PRIMARY OUTCOMES:
Fall risk | 10 minutes
  Balance - the body's ability to remain stable against internal and external factors.Clinical, Functional and computer aided methods are frequently used to evaluate balance. The risk of falling will be evaluated with the computerized static posturography device [Tetrax® Interactive Postural Balance System (Sunlight Medical, Israel)]
Fall risc | 5 minutes
  Balance - the body's ability to remain stable against internal and external factors.Clinical, Functional and computer aided methods are frequently used to evaluate balance. The risk of falling will be evaluated with the timed up to go test.

SECONDARY OUTCOMES:
Plantar Pressure Analysis | 10 minutes
  Static foot pressure measurement will be performed with (Emed, Novel GmBH,Germany)
  device in all cases.Peak pressure (Kpa), maximum force (N) and total foot area (cm²) values will be obtained.The correlation of these parameters with the risk of falling will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Shahla Alimadatli, Principal Investigator — Istanbul University - Cerrahpasa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Michaudet C, Edenfield KM, Nicolette GW, Carek PJ. Foot and Ankle Conditions: Pes Planus. FP Essent. 2018 Feb;465:18-23. PMID 29381041
- [Background] Cote KP, Brunet ME, Gansneder BM, Shultz SJ. Effects of Pronated and Supinated Foot Postures on Static and Dynamic Postural Stability. J Athl Train. 2005 Mar;40(1):41-46. PMID 15902323
- [Background] Knapp PW, Constant D. Posterior Tibial Tendon Dysfunction. 2024 May 21. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK542160/ PMID 31194317
- [Background] Mosca VS. Flexible flatfoot in children and adolescents. J Child Orthop. 2010 Apr;4(2):107-21. doi: 10.1007/s11832-010-0239-9. Epub 2010 Feb 18. PMID 21455468
- [Background] Forriol F, Pascual J. Footprint analysis between three and seventeen years of age. Foot Ankle. 1990 Oct;11(2):101-4. doi: 10.1177/107110079001100208. PMID 2265808
- [Background] Staheli LT, Chew DE, Corbett M. The longitudinal arch. A survey of eight hundred and eighty-two feet in normal children and adults. J Bone Joint Surg Am. 1987 Mar;69(3):426-8. PMID 3818704
- [Background] Awale A, Hagedorn TJ, Dufour AB, Menz HB, Casey VA, Hannan MT. Foot Function, Foot Pain, and Falls in Older Adults: The Framingham Foot Study. Gerontology. 2017;63(4):318-324. doi: 10.1159/000475710. Epub 2017 May 9. PMID 28482340
- [Background] Neri SGR, Harvey LA, Tiedemann A, Gadelha AB, Lima RM. Obesity and falls in older women: Mediating effects of muscle quality, foot loads and postural control. Gait Posture. 2020 Mar;77:138-143. doi: 10.1016/j.gaitpost.2020.01.025. Epub 2020 Feb 1. PMID 32036318
- [Background] Skopljak A, Muftic M, Sukalo A, Masic I, Zunic L. Pedobarography in diagnosis and clinical application. Acta Inform Med. 2014 Dec;22(6):374-8. doi: 10.5455/aim.2014.22.374-378. Epub 2014 Dec 19. PMID 25684844
- [Background] Akkaya N, Doganlar N, Celik E, Aysse SE, Akkaya S, Gungor HR, Sahin F. TEST-RETEST RELIABILITY OF TETRAX(R) STATIC POSTUROGRAPHY SYSTEM IN YOUNG ADULTS WITH LOW PHYSICAL ACTIVITY LEVEL. Int J Sports Phys Ther. 2015 Nov;10(6):893-900. PMID 26618068